CLINICAL TRIAL: NCT02393235
Title: A Comparative Analysis of Ovarian, Uterine and Spiral Arterial Blood Flow in Unexplained Infertility, Tubal Infertility and Fertile Groups
Brief Title: A Comparative Analysis of Arterial Blood Flow in Unexplained Infertility, Tubal Infertility and Fertile Groups
Status: Completed | Type: Observational
Sponsor: Suleymaniye Birth And Women's Health Education And Research Hospital (Other Government)
Collaborators: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AGZ1-UN-DOP
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
Keywords: unexplained infertility; tubal infertility; pulsatility index; resistance index; fertile women
MeSH Terms: conditions — Infertility | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- unexplained infertility(n:75): Ovarian, uterine and spiral artery pulsatility index and resistance index will measure with doppler ultrasonography in the mid-luteal phase. ( 21th day)
  Interventions: Other: doppler ultrasonography
- tubal infertility(n:75): Ovarian, uterine and spiral artery pulsatility index and resistance index will measure with doppler ultrasonography in the mid-luteal phase. ( 21th day)
  Interventions: Other: doppler ultrasonography
- fertile group(n:75): Ovarian, uterine and spiral artery pulsatility index and resistance index will measure with doppler ultrasonography in the mid-luteal phase. ( 21th day)
  Interventions: Other: doppler ultrasonography

INTERVENTIONS:
Other: doppler ultrasonography — Ovarian, uterine and spiral artery pulsatility index and resistance index will measure

SUMMARY:
Factors affecting the success of the treatment of infertility can evaluate before and after embryo transfer in two stages. Most of the patients reach the embryo transfer stage. Unfortunately, the investigators are able to intervene very few of the factors that will affect the success of the post-transfer. All factors and treatments that affect the implantation is vital to identify. Basically, healthy vasculature is essential for a successful implantation. The investigators will try to understand relationship between vascular resistance and type of infertility. The investigators will examine whether the effect of the ovarian uterine and spiral artery resistance over infertility.

DETAILED DESCRIPTION:
In this study the investigators will examine whether the alterations of doppler indices in the uterine, ovarian and spiral arteries can help to explain tubal or unexplained infertility as a standard screening method. Patients in unexplained-tubal infertility groups were treated in our IVF clinic. Patients will be invited to the hospital according to the criteria of the study. Fertile patients will be selected according to the criteria for patients who have come for the annual smear control. The study hypothesis is that the resistance in ovarian, uterine and spiral artery doppler will be higher in cases with tubal and unexplained infertility as opposed to low resistance in fertile women.Ovarian, uterine and spiral artery pulsatility index (PI = (peak systolic velocity - end diastolic velocity) / time averaged velocity and resistance index ( RI= (peak systolic velocity - end diastolic velocity) / peak systolic velocity ) will measure with doppler ultrasonography in the mid-luteal phase ( 21th day). Measured values are to be compared.

ELIGIBILITY:
Inclusion Criteria:

* unsuccessful infertility treatment
* normal prolactin levels
* normal thyroid stimulation hormone levels
* no ovarian or pelvic surgery history

Exclusion Criteria:

* To have systemic diseases
* receive medical treatments which may influence the clearance or excretion of gonadotropins and sex steroids

Ages: 22 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women received infertility treatment
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study is to evaluate the possible difference in ovarian artery impedance to blood flow ( RI and PI) among unexplained infertility, tubal infertility and fertile group. | 2-3 month
The primary outcome measure of this study is to evaluate the possible difference in uterine artery impedance to blood flow (RI and PI) among unexplained infertility, tubal infertility and fertile group. | 2-3 month
The primary outcome measure of this study is to evaluate the possible difference in spiral artery impedance to blood flow ( RI and PI) among unexplained infertility, tubal infertility and fertile group. | 2-3 month

CONTACTS AND LOCATIONS:
Overall Officials: Ali G Zebitay, M.D., Principal Investigator — Suleymaniye Birth And Women's Health Education And Research Hospital
Locations (1):
- Suleymaniye Birth And Women's Health Education And Research Hospital, Istanbul, Turkey (Türkiye)